CLINICAL TRIAL: NCT01808833
Title: A Pilot Trial of Frailty Assessment in Older Adults (Age 70 >) Requiring Concurrent Chemotherapy Plus Radiation Therapy for Cancer (CTRC# 12-22)
Brief Title: Frailty Study of Older Adults Getting Chemotherapy and Radiation Therapy
Status: Terminated | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: CTRC 12-22
Record Dates: First submitted 2012-11-01; First posted 2013-03-11 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Cancer
Keywords: Frailty; Geriatric oncology
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Frail patients
- Non-frail patients

SUMMARY:
The investigators hypothesize that frailty assessment prior to concurrent chemotherapy and radiation therapy in the elderly will predict treatment-related toxicity and morbidity and that such assessment at serial time points will help improve treatment and outcomes for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following histologically or cytologically confirmed cancers: lung cancer, head and neck cancer, gastric cancer, anal cancer, rectal cancer, cervix cancer, or bladder cancer, and must have appropriate indications for the use of standard concurrent chemotherapy plus radiation therapy as defined in the NCCN (National Comprehensive Cancer Network) Guidelines for each of these specific organ-sites.
* Age >70 years.
* ECOG (Easter Cooperative Oncology Group) performance status of 0, 1 or 2.
* Life expectancy Tables showing upper, middle, and lower quartiles of life expectancy for women and men age 70 and older should be used and life expectancy should be estimated to be of sufficient to justify the use of concurrent chemotherapy plus radiation for each organ site and indication.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered to baseline from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any investigational agents.
* Patients with known distant site metastases (M1 disease) or brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have a history of one or more other concurrent cancers besides the cancer for which concurrent chemotherapy plus radiation therapy is considered are ineligible only if the other cancer or cancers are being considered for treatment or are actively being treated.
* Patients carrying a pre-existing diagnosis of HIV/AIDS and are on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with chemotherapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with any standard contraindication to chemotherapy or radiation therapy are ineligible.
* Transplant recipient patients on immune-suppressant agents are ineligible due to increased risk of infection.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Age >70 years undergoing concurrent standard of care chemotherapy plus radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in frailty assessment due chemotherapy toxicity | Subjects will be followed for frailty measures during standard of care chemotherapy treatment, an average of 8 weeks per treatment
  Validated frailty measures, and geriatric assessment tools will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Karnad, MD, Principal Investigator — University of Texas
Locations (1):
- Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States